CLINICAL TRIAL: NCT03153033
Title: The Effect of a Wheelchair Propulsion-induced Fatigue Protocol on Biomechanical and Neuromuscular Risk Factors of Shoulder Pain in Persons With a Spinal Cord Injury Living in Switzerland: a Cross-sectional Study With a Repeated Measures Within Subject Design
Brief Title: Fatigue Induced by Overground Wheelchair Propulsion in Persons With a Spinal Cord Injury: Upper Limb Saving or Straining?
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Collaborators: Human Engineering Research Laboratories (Other); University Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-13
Record Dates: First submitted 2017-05-04; First posted 2017-05-15 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Spinal Cord Injuries; Fatigue; Muscle, Heart
Keywords: Wheelchair propulsion; Shoulder; Biomechanics
MeSH Terms: conditions — Spinal Cord Injuries; Fatigue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Fatigue protocol — The figure 8 protocol (fatigue intervention) requires the participants to propel three times as many laps as possible for four minutes each with their wheelchair. The protocol has been developed and used previously. Every bout of four minutes is separated by 90 seconds of rest. Each lap consists of a right and left turn and two complete stops after half a lap. Measurements during the protocol include the Rate of Perceived Exertion (RPE) scale, heart rate, and propulsion kinetics.

SUMMARY:
What are the implications of wheelchair propulsion-induced fatigue for the development of shoulder pain and how can this knowledge improve prevention programs?

With this project, the "Shoulder Health and Mobility group" of the Swiss Paraplegic Research in Nottwil (Switzerland) wants to investigate how fatigue during wheelchair propulsion affects risk factors for shoulder pain of persons with a spinal cord injury (SCI). The investigators want to find out how the handrim wheelchair propulsion technique changes with fatigue and want to define persons who are susceptible to fatigue.

Getting life back after a SCI will most likely occur with the help of a wheelchair, whether it is at the beginning of rehabilitation or throughout further life. Gaining back mobility and participation in social life is important, also because of the multiple positive effects of physical activity on person's health and self-esteem, preventing several chronic diseases. Therefore, it is needed to try to stay away from shoulder injuries. Since the shoulder is very mobile and thus unstable, the joint is at increased risk for injuries. This is reflected in the high amount of persons with a SCI having shoulder pain (between 30 to 70 %). Once pain or an injury occurred, it is hard to recover, as so far no effective treatment is available. Several factors as gender, weight, age, level and completeness of the SCI, movement patterns and muscle strength were found to be related with injury and pain. However, it is currently not well understood what exactly causes shoulder injuries.

Handrim wheelchair propulsion is an inefficient mode of propulsion and asks a lot of demands to the upper body. Because of the inefficient movement and the shoulder being prone to injuries, wheelchair propulsion has a high chance of inducing shoulder injuries and pain. Propelling with a technique minimizing the loads on the shoulders and improving the capacity to perform these movements (as increasing muscle strength) is of utmost importance as these factors can be modified by training. Previous intervention programs have learned wheelchair users to propel with long and smooth strokes aiming to reduce the loads. Although someone might be aware of the recommended techniques and can apply them, propulsion technique might change with fatigue and could become less optimal. A similar phenomena happens for example in landing strategies from a jump. In a fresh state, persons will try to have a stable landing reducing the impact on the lower limbs. With fatigue, however, there will be a tendency to forget about the proper landing technique which on its turn can increase the risk of injuries. This was suggested to be one of the reasons why there is an increased prevalence of injuries towards the end of a game. So far, it is unclear how fatigue alters propulsion technique and how these changes are related with an increased risk of shoulder pain.

Tis project aims to achieve the goals by investigating how very strenuous wheelchair propulsion (fatigue intervention) of 15 minutes alters the propulsion technique of 50 persons with a SCI. All participants will perform the fatigue protocol in the movement analysis lab at the Swiss Paraplegic Research. During the protocol, participants will be requested to perform as many 8 loops as possible with their wheelchairs, including starts, stops, and right and left turns. Before and after the protocol, movement patterns, muscle usage and loads during wheelchair propulsion and the characteristics of the shoulder muscle tendons during rest will be assessed. Furthermore, the person's characteristics, such as weight, age, gender, time since injury, injury level, health conditions, use of medication, muscle strength and activity levels will be assessed. All these factors might be associated with the susceptibility to fatigue.

To answer our questions, we will first compare the propulsion technique (movement patterns, loads, and muscle usage) before and after the protocol to investigate the direct effect of fatigue. Secondly, we will investigate the association of negative changes in tendon appearance (which has been related to injury) with the changes in the propulsion technique to investigate the implications of acute changes that might increase the risk of injury. Finally we will run a model including all variables to determine which person's characteristics are associated with an increased susceptibility to fatigue.

The results will be highly relevant as it will give answers about the content, the aims and the target population of prevention programs for shoulder injury, aiming to improve mobility, participation, and quality of life in persons with SCI.

DETAILED DESCRIPTION:
Background and rationale:

Wheelchairs are the most important assistive devices used by persons with a spinal cord injury (SCI). A Danish study reported for example that 83.5% of 236 persons used a manual wheelchair and 27% a powered wheelchair, some of which used both a manual and an electrical wheelchair. The repetitive nature of wheelchair propulsion in combination with the shoulder being prone to injuries results in a high prevalence of persons with a SCI having shoulder pain. Several factors have been associated with shoulder pain but exact pathways remain unclear. In order to improve injury prevention which would have a significant effect on shoulder pain, it is important to focus on biomechanical and neuromuscular risk factors modifiable by training. Fatigue could have a negative effect on propulsion mechanics further increasing the risk of injury. Previous studies have induced fatigue by interventions on a treadmill or with an ergometer. However, it is important to investigate functional fatigue, as the effect of fatigue is task dependent. To date there is no clear understanding of the effect of functional fatigue on biomechanical and neuromuscular risk factors in persons with SCI during wheelchair propulsion.

Objectives:

Main objective: What is the role of muscle fatigue in altering neuromusculoskeletal and movement body functions and structures related to shoulder pain in persons with SCI? Aim1: To define how muscle fatigue induced by wheelchair propulsion changes biomechanical and neuromuscular risk factors of shoulder injuries, leading to shoulder pain, in persons with SCI.

Aim 2: To evaluate how changes in propulsion biomechanics due to propulsion-induced fatigue are associated with changes in tendon appearance related to tendinopathy, in persons with SCI.

Aim 3: To identify predictor variables (e.g., activity levels and muscle strength) for persons with SCI who are susceptible to wheelchair propulsion-induced fatigue.

Study design: Repeated measures within subject design

For this study, 50 participants will be recruited via the Swiss Spinal Cord Injury Cohort study database. The number of 48 participants was calculated based on a sample-size estimation from a study investigating a high-intensity wheelchair propulsion activity that found that echogenicity ratio changed significantly from 1.97 ± 0.74 to 1.73 ± 0.56 (p=0.038) (after the intense wheelchair propulsion activity. To observe this change of 0.24 difference in echogenicity ratio of the biceps tendon at 80% statistical power and alpha=0.05, 48 participants are needed. In order to take into account drop-out and missing data 50 participants will be recruited. All participants will meet the defined inclusion criteria and excluded when meeting the exclusion criteria.

Data collection:

Participants will be tested during one session of four hours after they have read and signed the informed consent. During the testing session the following measurements will be performed:

Participant's characteristics and activity levels: Socio-demographic variables, injury characteristics, presence of contractures and spasticity will be defined with a general questionnaire. Furthermore, activity levels will be defined with the Physical Activity Scale for Individuals with Physical Disabilities (PASIPD).

Participants weight will be measured.

Quantitative ultrasound pre-fatigue: Ultrasound measurements of the biceps brachii and supraspinatus tendon at rest will be collected with Quantitative Ultrasound Protocols (QUS). This technique has been used previously and has proven strong reliability and validity for measures of shoulder pain and tendinopathy. More specifically, for the biceps tendon longitudinal image, participants will be positioned with their non-dominant arm flexed 90˚ at the elbow and their wrist resting on the ipsilateral thigh. Images will be taken so that the fibres are aligned perpendicular to the transducer which optimises the quantification of fibre alignment and tendon thickness. In order to mark the skin location of the pre-fatigue measurement, a steel reference marker will be taped to the skin at the distal end of the transducer. The distinct interference pattern created by the marker at the top of the images is used to define the region of interest (ROI) upon which the computations are performed. For the supraspinatus transverse image, participants will be positioned with their non-dominant palm placed on the lower back, shoulder extended, and elbow flexed posteriorly. The steel marker is now taped to the skin at the proximal end of the transducer and the widest part of the tendon is imaged. The specific positions optimize image quality and repeatability of the imaging protocol. Furthermore, three consecutive measurements of the acromio-humeral distance of the non-dominant hand will be collected under an unloaded and loaded conditions (during push up in wheelchair, once without further instructions and once with the instruction of retracting the shoulders) as has been done previously.

The same trained investigator will perform all ultrasound measurements.

Maximum sprint and strength test: A 15m over ground sprint test will be performed to define anaerobic work capacity. Furthermore a maximum isometric forward push against resistance on the wheelchair will be performed to measure maximal strength.These tests have been used previously. During both tests, external forces will be collected at 100 Hz with the SmartWheel. The 15m sprint aims to define the anaerobic work capacity. The participants will be required to propel as fast as possible from one cone to another standing 15 meters apart which will result in an outcome of the maximum unilateral power output. For the isometric maximum push, the wheelchair with SmartWheel will be connected via a rope to a force transducer and a wall. The participant will be requested to push as hard as possible for 5 seconds with the hands on top of the handrim to measure the maximum applied force.

Wheelchair propulsion pre-fatigue: The participant will be requested to propel his/her wheelchair on the treadmill for two trials of 90 seconds at two power output conditions (intermediate and hard). During the trials, 3D kinematics of the upper extremity, 3D kinetics applied to the handrim of the wheelchair and muscle activation of muscles active during wheelchair propulsion will be collected.

Fatigue protocol: The figure 8 protocol (fatigue intervention) requires the participants to propel three times as many laps as possible for four minutes each. Every bout of four minutes is separated by 90 seconds of rest. Each lap consists of a right and left turn and two complete stops after half a lap. Measurements during the protocol include the Rate of Perceived Exertion (RPE) scale, heart rate, and propulsion kinetics.

Wheelchair propulsion and Quantitative ultrasound post-fatigue: The same measurements as in the pre-fatigue tests will be performed.

Statistical considerations:

Aim 1: To investigate the effect of muscle fatigue induced by wheelchair propulsion on biomechanical and neuromuscular risk factors of shoulder injuries, leading to shoulder pain, in persons with SCI.

Hypothesis 1: Muscle fatigue induced by wheelchair propulsion will result in significant changes in biomechanical and neuromuscular risk factors related to shoulder pathology.

Dependent variables of interest are stroke frequency, glenohumeral contact force, net joint moments, kinematic and normalised muscle forces during wheelchair propulsion, tendon appearance of the m. biceps brachii and m. supraspinatus, and acromio-humeral distance. A statistical parametric mapping (SPM) one way repeated measures ANOVA will be used to assess meaningful variations across time for each continuous variable during wheelchair propulsion (alpha=0.05).

Aim 2: To determine the relation between changes in propulsion biomechanics and changes in tendon appearance related to tendinopathy post-fatigue, in persons with SCI.

Hypothesis 2: There will be a positive association between changes in propulsion biomechanics and changes in tendon appearance of the m.biceps and m.supraspinatus when controlling for sex, level and completeness of injury, health conditions, range of motion and weight.

Independent variables will be changes in propulsion biomechanics that significantly changed after the fatigue protocol and dependent variables will include changes in tendon appearance of the m.biceps and m.supraspinatus. Covariates will be sex, level and completeness of injury, health conditions (spasticity and contractures), range of motion and weight. Multivariable linear regression analysis will be used to test the hypothesis

Aim 3: To investigate the relation of the susceptibility of fatigue and person's characteristics (activity levels and muscle strength), in persons with SCI.

Hypothesis 3: There will be a negative association between changes in propulsion biomechanics (including stroke frequency, scapular kinematics and glenohumeral contact force) and both activity levels and muscle strength, when controlling for sex, level and completeness of injury, health conditions (spasticity and contractures), range of motion and weight.

Independent variables will be propulsion biomechanics that significantly changed after the fatigue protocol and dependent variables will include physical activity levels and muscle strength. Covariates will be sex, level and completeness of injury, health conditions (spasticity and contractures), range of motion and weight. Multivariable linear regression analysis will be used to test the hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults with non-progressive traumatic or non-traumatic SCI with permanent residence in Switzerland.
* Diagnosed with a paraplegia (lesion level T2-L1)
* At least 1 year post discharge from rehabilitation
* Use a handrim wheelchair for daily use and no required support for moving around for more than 100m with the handrim wheelchair
* Able to manually propel a wheelchair for at least 15 minutes continuously
* German or French speaking

Exclusion Criteria:

* New SCI in context of palliative care
* SCI due to congental conditions, neurodegenerative disorders, or Guillain-arré syndrome.
* Upper extremity pain that limits their ability to propel the wheelchair
* History of shoulder, elbow, or wrist fractures/dislocations that are still causing symptoms
* History of cardiopulmonary problems that could be exacerbated by strenuous physical activity
* The wheelchair has no quick release axle

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will investigate healthy individuals with a SCI. Suitable participants will be identified based on the SwiSCI community survey (EKNZ registration number 1008). Suitable persons will be selected based on age (18-65 years), lesion level of SCI (paraplegia), language (German and French), time since injury, and use of wheelchair for daily activities. These persons will be contacted by letter and asked whether they are interested in participating in the study. After initial screening, further selection will be done using a questionnaire and further contact will be done by either telephone, e-mail or written letter (participants preference).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Echogenicity ratio of the biceps brachii tendon | 4 hours
  This is the ratio of the tendon pixel grayscale and the muscle pixel grayscale of the muscle above the tendon.

SECONDARY OUTCOMES:
Shoulder load | 4 hours
  Defined as the glenohumeral contact force (3D total force of the head of the humerus against the glenoid fossa). This outcome will be based on a computerized model that uses kinetic and kinematic data. An instrumented wheelchair wheel will provide the kinetic data. The kinematic data will be measured with an eight-camera infrared camera system, using passive markers. In wheelchair research, this is the most widely accepted way of collecting data, since it is non-invasive as well as accurate.
Shoulder kinematics | 4 hours
  The shoulder kinematics will be defined as the relative orientations of the bony segments of the shoulder (thorax, clavicle, scapula and humerus) in 3D. The calculations will be done in agreement with the ISB definitions. The data will be provided with an eight-camera infrared camera system, using reflective markers.
Contact time | 4 hours
  This is the amount of time that the hand spends on the push rim during a stroke of wheelchair propulsion. An instrumented wheelchair wheel will provide the kinetic data from which contact time can be calculated.
Muscle activity patterns of the biceps brachii | 4 hours
  Muscular activation of the biceps brachii will be identified during the push phase of treadmill wheelchair propulsion.
Muscle activity patterns of the upper trapezius | 4 hours
  Muscular activation of the upper trapezius will be identified during the push phase of treadmill wheelchair propulsion.
Muscle activity patterns of the lower trapezius | 4 hours
  Muscular activation of the lower trapezius will be identified during the push phase of treadmill wheelchair propulsion.
Muscle activity patterns of the deltoideus | 4 hours
  Muscular activation of the deltoideus will be identified during the push phase of treadmill wheelchair propulsion.
Muscle activity patterns of the pectoralis major | 4 hours
  Muscular activation of the pectoralis major will be identified during the push phase of treadmill wheelchair propulsion.

OTHER OUTCOMES:
sex | 10 minutes
  This is the biological sex of the participant
Activity levels | 20 minutes
  will be defined with a valid questionnaire (Physical Activity Scale for Individuals with a Disability (PASIPD)) at the beginning of data-collection to reduce recall-bias.
Weight | 15 minutes
  Weight of the person will be defined as the weight of the participant and the wheelchair minus the weight of the wheelchair itself.
Sprint time | 2 hours
  Duration of a 15 m overground wheelchair propulsion sprint test.
Maximum power output | 2 hours
  Maximum power output of an isometric push against resistance.
Etiology of the spinal cord injury | 10 minutes
  The participant will be asked whether the spinal cord injury has a traumatic or non-traumatic etiology
Lesion level of the spinal cord injury | 10 minutes
  The participant will be asked for the lesion level of the spinal cord injury (e.g., Thoracic 7-8).
Completeness of the spinal cinjury | 10 minutes
  The participant will be asked whether the spinal cord injury is complete or incomplete.
Time since injury of the spinal cord injury | 10 minutes
  The time since injury will be calculated from the data of measurement and the date the spinal cord injury occurred.
Health condition spasticity | 10 minutes
  Spasticity in the upper extremities will be reported via questions that will be asked to the persons.
Health condition contractures | 10 minutes
  Contractures in the upper extremities will be reported via questions that will be asked to the persons.

CONTACTS AND LOCATIONS:
Overall Officials: Fransiska Marie Bossuyt, Msc, Principal Investigator — Swiss Paraplegic Research, Nottwil
Locations (1):
- Swiss Paraplegic Research, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mackenzie TA, Bdaiwi AH, Herrington L, Cools A. Inter-rater Reliability of Real-Time Ultrasound to Measure Acromiohumeral Distance. PM R. 2016 Jul;8(7):629-34. doi: 10.1016/j.pmrj.2015.11.004. Epub 2015 Nov 19. PMID 26603199
- [Result] Collinger JL, Gagnon D, Jacobson J, Impink BG, Boninger ML. Reliability of quantitative ultrasound measures of the biceps and supraspinatus tendons. Acad Radiol. 2009 Nov;16(11):1424-32. doi: 10.1016/j.acra.2009.05.001. Epub 2009 Jul 10. PMID 19596592
- [Result] Biering-Sorensen F, Hansen RB, Biering-Sorensen J. Mobility aids and transport possibilities 10-45 years after spinal cord injury. Spinal Cord. 2004 Dec;42(12):699-706. doi: 10.1038/sj.sc.3101649. PMID 15289807
- [Result] Enoka RM, Duchateau J. Translating Fatigue to Human Performance. Med Sci Sports Exerc. 2016 Nov;48(11):2228-2238. doi: 10.1249/MSS.0000000000000929. PMID 27015386
- [Result] Collinger JL, Impink BG, Ozawa H, Boninger ML. Effect of an intense wheelchair propulsion task on quantitative ultrasound of shoulder tendons. PM R. 2010 Oct;2(10):920-5. doi: 10.1016/j.pmrj.2010.06.007. PMID 20970761
- [Result] van Drongelen S, Boninger ML, Impink BG, Khalaf T. Ultrasound imaging of acute biceps tendon changes after wheelchair sports. Arch Phys Med Rehabil. 2007 Mar;88(3):381-5. doi: 10.1016/j.apmr.2006.11.024. PMID 17321833
- [Result] van der Scheer JW, de Groot S, Tepper M, Gobets D, Veeger DH; ALLRISC group; van der Woude LH. Wheelchair-specific fitness of inactive people with long-term spinal cord injury. J Rehabil Med. 2015 Apr;47(4):330-7. doi: 10.2340/16501977-1934. PMID 25594246
- [Result] van der Helm FC. A finite element musculoskeletal model of the shoulder mechanism. J Biomech. 1994 May;27(5):551-69. doi: 10.1016/0021-9290(94)90065-5. PMID 8027090
- [Result] van der Helm FCT. A thee dimensional model of the shoulder and elbow. First conference of the international shoulder group. Shaker Publishers BV, Delft University of Technology, The Netherlands. 1997.
- [Derived] Minder U, Arnet U, Muller E, Boninger M, Bossuyt FM. Changes in neuromuscular activation, heart rate and rate of perceived exertion over the course of a wheelchair propulsion fatigue protocol. Front Physiol. 2023 Oct 18;14:1220969. doi: 10.3389/fphys.2023.1220969. eCollection 2023. PMID 37920802